CLINICAL TRIAL: NCT02024321
Title: Phase 1: Select Tumor Patients to be Observed Phase 2: Observe the Blood Glucose Values During TPN Phase 3: Sort Data
Brief Title: Study on Blood Glucose Variations in Tumor Patients Before and After Total Parenteral Nutrition
Acronym: TPN
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jincheng Yang, pharmacist, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: TPN-tumor
Record Dates: First submitted 2013-12-18; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Cancer; Surgery; Nutrition Related Cancer
Keywords: abdominal surgery; TPN; blood glucose
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tumor patients, TPN, surgery: This work involved prospective study of surgical patients receiving TPN during the calendar year of 2013 at Cancer Hospital.

SUMMARY:
The purpose of this study is to determine the relationship among TPN, tumor and blood glucose.

DETAILED DESCRIPTION:
Select the tumor patients in abdominal department after surgery with TPN. Monitor the blood glucose variation after TPN.

ELIGIBILITY:
Inclusion Criteria:

* 1.tumor patients,2.use TPN after surgery

Exclusion Criteria:

* without using TPN

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tumor patients using TPN in abdominal surgery department in Cancer Hospital.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Glycemic Variations during TPN | 1 year
  Observe the blood glucose variation in tumor patients after surgery. According to the TPN infusion time, the blood glucose values are divided into three parts: pre TPN, within 24h and after 24h.

CONTACTS AND LOCATIONS:
Overall Officials: Jincheng Yang, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Pasquel FJ, Spiegelman R, McCauley M, Smiley D, Umpierrez D, Johnson R, Rhee M, Gatcliffe C, Lin E, Umpierrez E, Peng L, Umpierrez GE. Hyperglycemia during total parenteral nutrition: an important marker of poor outcome and mortality in hospitalized patients. Diabetes Care. 2010 Apr;33(4):739-41. doi: 10.2337/dc09-1748. Epub 2009 Dec 29. PMID 20040658
- [Derived] Yang JC, Dai YY, Wang LM, Xie YB, Zhou HY, Li GH. Glycemic Variation in Tumor Patients with Total Parenteral Nutrition. Chin Med J (Engl). 2015 Aug 5;128(15):2034-9. doi: 10.4103/0366-6999.161358. PMID 26228214